CLINICAL TRIAL: NCT02920801
Title: Study About Effect of Saxagliptin on Circulating Endothelial Progenitor Cells and Endothelial Function in Newly Diagnosed Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Yan Ling, associate professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13040490434
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: saxagliptin; endothelial progenitor cell; flow-mediated dilation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

ARMS (2):
- saxagliptin group (Experimental): saxagliptin group consumed saxagliptin 5mg per day for 12 week
  Interventions: Drug: saxagliptin
- metformin group (Active Comparator): metformin group consumed metformin 1500mg per day for 12 week
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: saxagliptin — 5mg per day for 12 weeks
  Arms: saxagliptin group
Drug: Metformin — 1500mg per day for 12 weeks
  Arms: metformin group

SUMMARY:
In this study, the investigators aim to investigate whether saxagliptin modulate endothelial progenitor cells number and flow-mediated dilation in newly diagnosed, treatment-naive type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetics (diagnosis were made according to the American Diabetes Association Guideline [19] ), treatment naive, age 30-75, hemoglobin A1c (HbA1c) ≥6.5%, fasting c-peptide >1.0ng/L

Exclusion Criteria:

* pregnancy or lactation, smoker, acute disease or infection, chronic renal disease (estimated glomerular filtration rate <60 mL/min/1.73m2), live enzymes 3 times above the normal range, positive islet autoantibody, fasting c-peptide <1.0ng/L, severe hypertriglyceridemia (triglyceride >5.6mmol/L), cardiovascular events or surgery within 3 months, taking glucocorticoid, history of acute or chronic pancreatitis, pancreatic tumor, severe cardiac or pneumonic disease.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
endothelial progenitor cell | 12weeks
flow-mediated dilation | 12weeks

SECONDARY OUTCOMES:
HbA1c | 12weeks
fasting blood glucose | 12weeks
2 hour postprandial blood glucose | 12weeks
liver function test | 12weeks
renal function test | 12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Li, Shanghai, Shanghai Municipality, China